CLINICAL TRIAL: NCT02763072
Title: A Single-Center 2-Arm Study of the Enlighten and Excel V Laser for Lentigines on the Hands
Brief Title: A Single-Center 2-Arm Study for Lentigines on the Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-16-EV09
Record Dates: First submitted 2016-04-25; First posted 2016-05-05 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Lentigines
MeSH Terms: conditions — Lentigo

STUDY DESIGN:
Oversight: FDA-regulated Device: Yes

ARMS (2):
- Enlighten Laser (Experimental): 12 subjects will receive treatment the Enlighten laser.
  Interventions: Device: Enlighten Laser
- Excel V Laser (Active Comparator): 12 subjects will receive treatment with the Excel V laser.
  Interventions: Device: Excel V Laser

INTERVENTIONS:
Device: Enlighten Laser
  Arms: Enlighten Laser
Device: Excel V Laser
  Arms: Excel V Laser

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of two laser systems for improvement of lentigines on the hands.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness and safety in a clinic setting of two laser systems for the treatment of lentigines (liver spots, age spots, or dark sun spots) on the hands.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, 30-90 years of age (inclusive).
2. Fitzpatrick Skin Type I - III.
3. Desires non-invasive and non-ablative treatment of lentigines on the hand(s).
4. Have 4 or more lentigines on the hand(s).
5. Subject must be able to read, understand and sign the Informed Consent Form.
6. Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
7. Willing to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treatment area every day for the duration of the study, including the follow-up period.
8. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
9. Agree to not undergo any other procedure(s) for treatment of lentigines during the study, including but not limited to chemical peel, laser and light based device treatment, and home-use device treatment.
10. Agree to not undergo any injection of botulinum toxin, collagen, hyaluronic acid filler or other dermal filler to the treatment area during the study.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug in the target area within 6 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation, such as laser or light-based procedures or surgery.
3. Systemic use of retinoid, such as isotretinoin, within 6 months of study participation.
4. Use of topical medications on the hands, such as antibiotics, benzoyl peroxide, retinoids (isotretinoin), corticosteroids, hydroquinone, or products containing dihydroxyacetone or alpha-hydroxy with concentration > 8%, within 1 month of participation.
5. History of malignant tumors in the target area.
6. Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles.
7. Pregnant.
8. Having an infection, dermatitis, or a rash in the treatment area.
9. History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
10. Any use of medication that is known to increase sensitivity to light according to investigator's discretion.
11. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
12. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
13. Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
14. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
15. In the opinion of the investigator, any physical or mental condition which might make it unsafe for the subject to participate in this study or which requires systematic therapy that could interfere with this research study.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Stankiewicz, MD FAAD, Principal Investigator — DuPage Medical Group
Locations (1):
- DuPage Medical Group, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Excel V Laser: 12 subjects will be enrolled in the Excel V group, .
- Enlighten Laser: 12 subjects will be enrolled in the Enligthen group
Period: Overall Study
Arm/Group | Excel V Laser | Enlighten Laser
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Excel V Laser: 12 subjects will be enrolled in the Excel V group
- Enlighten Laser: 12 subjects will be enrolled in the Enlighten group
- Total: Total of all reporting groups
Arm/Group | Excel V Laser | Enlighten Laser | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0) | 64.8 (8.6) | 63.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in the Number of Hand Lentigines as Assessed by Blinded Reviewers.
Time Frame: 4 weeks post-final treatment
Population: Study terminated prior to outcome data collected due to company change in priorities.
Groups:
- Enlighten Laser: 12 subjects will receive treatment with the Enlighten laser.
Arm/Group | Enlighten Laser | Excel V Laser
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Physician's Global Assessment Score of the Overall Appearance of the Hands
Description: Degree of improvement in the overall appearance of the hands as assessed by blinded reviewers using the Physician's Global Assessment scale: 4=Very Significant Improvement,3=Significant Improvement, 2=Moderate Improvement, 1=Mild Improvement and 0=No Change Higher scores indicate better outcomes
Time Frame: 4 weeks post final treatment
Population: 1 subject was lost to follow up in the Excel V group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enlighten Laser | Excel V Laser
Number analyzed (Participants) | 12 | 11
score on a scale | 3.8 (0.6) | 3.9 (0.3)

3. Secondary Outcome: Physician's Global Assessment Score of Skin Texture of the Hands
Description: Degree of improvement in the Skin Texture of the hands as assessed using the Physician's Global Assessment scale: 4=Very Significant Improvement,3=Significant Improvement, 2=Moderate Improvement, 1=Mild Improvement and 0=No Change. Higher scores indicate better outcomes
Time Frame: 4 weeks post final treatment
Population: 1 subject was lost to follow up in the Excel V group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enlighten Laser | Excel V Laser
Number analyzed (Participants) | 12 | 11
score on a scale | 2.9 (1.8) | 3.1 (1.1)

4. Secondary Outcome: Subject Satisfaction
Description: Subject-completed questionnaire to rate their level of satisfaction with the laser treatment outcome
Time Frame: 4 weeks post final treatment
Population: 1 subject was lost to follow up in the Excel V group
Measure: Count of Participants; unit: Participants
Arm/Group | Enlighten Laser | Excel V Laser
Number analyzed (Participants) | 12 | 11
Participants
  Very Satisfied | 9 | 8
  Satisfied | 2 | 3
  Neutral | 1 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks post final treatment, up to 17 weeks
Arm/Group | Excel V Laser | Enlighten Laser
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Excel V Laser (N=12) | Enlighten Laser (N=12)
Erythema (Skin and subcutaneous tissue disorders) | 6 | 9
Darkening of vessel (Skin and subcutaneous tissue disorders) | 0 | 5
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT02763072/Prot_SAP_000.pdf